CLINICAL TRIAL: NCT06688994
Title: Vitamin D Metabolites as Biomarkers for the Identification of Kidney Injury in Cardiac Surgery
Acronym: VITAL
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 23-6027
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Acute Kidney Injuries; Chronic Renal Diseases
Keywords: Chronic renal disease; Acute kidney injury; Vitamin D
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators will be measuring vitamin D metabolites in blood samples drawn from patients undergoing cardiac surgery to determine the correlation with renal function as assessed by serum creatinine. The investigators will include 20 patients in each of the following 3 groups based on serum creatinine measured within 28-days of surgery: 1) normal kidney function (eGFR > 60 mL/min, n=20), 2) moderate impaired kidney function, eGFR between 30 and 60 mL/min (n=20) and 3) severe kidney dysfunction eGFR < 30 mL/min (n=20).

ELIGIBILITY:
Inclusion Criteria

* ≥ 18 years
* Patients undergoing cardiac surgery
* Serum Creatinine measured with 28 days of surgery

Exclusion Criteria

* Exogeneous calcitriol (1,25(OH)2D3) intake
* History of parathyroidectomy
* Patients with liver or kidney cancer
* Patients with liver disease (e.g. liver failure, cirrhosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery .
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine the correlation between eGFR as determined serum creatinine and vitamin D metabolites as markers of kidney function | Up to 1 month before surgery up until POD 7
  serum creatinine (sCr) and vitamin D metabolites (specifically 25(OH)D3 and 1,25(OH)2D3) will be measured in the same blood sample to determine the incidence of AKI and CKD in patients undergoing cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A McCluskey, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network-Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Data from this study is unique to the study and analytical techniques used

REFERENCES:
- [Result] Chow EC, Quach HP, Vieth R, Pang KS. Temporal changes in tissue 1alpha,25-dihydroxyvitamin D3, vitamin D receptor target genes, and calcium and PTH levels after 1,25(OH)2D3 treatment in mice. Am J Physiol Endocrinol Metab. 2013 May 1;304(9):E977-89. doi: 10.1152/ajpendo.00489.2012. Epub 2013 Mar 12. PMID 23482451
- [Result] Chow EC, Sondervan M, Jin C, Groothuis GM, Pang KS. Comparative effects of doxercalciferol (1alpha-hydroxyvitamin D(2)) versus calcitriol (1alpha,25-dihydroxyvitamin D(3)) on the expression of transporters and enzymes in the rat in vivo. J Pharm Sci. 2011 Apr;100(4):1594-604. doi: 10.1002/jps.22366. Epub 2010 Oct 21. PMID 20967888